CLINICAL TRIAL: NCT04324515
Title: Pilot Open Randomized Controlled Trial Comparing Patients Undergoing Robotic Gastric Bypass With or Without Concomitant Cholecystectomy
Brief Title: Randomized Trial Comparing Gastric Bypass With and Without Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Jung Minoa, Dr.med., University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-01243
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Roux-en-Y Gastric Bypass; Cholecystitis; Gallstone; Gallbladder Diseases
MeSH Terms: conditions — Cholecystitis; Gallstones; Gallbladder Diseases | interventions — Cholecystectomy

STUDY DESIGN:
Intervention Model Description: Patients who meet the inclusion criteria will be randomized according to a randomization list generated by the CRC of the University Hospital of Geneva. The randomization envelops will be opened by the study staff at the appropriate time prior to the scheduling of gastric bypass after subject selection. The randomization assignment insert will contain information specifying whether the cholecystectomy will be performed or not during gastric bypass procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arm without cholecystectomy (Other): Study Arm: Patients with gastric bypass without concomitant cholecystectomy
  Interventions: Procedure: Robotic gastric bypass with or without cholecystectomy
- Control Arm with cholecystectomy (Other): Control Arm: Patients with gastric bypass with concomitant cholecystectomy
  Interventions: Procedure: Robotic gastric bypass with or without cholecystectomy

INTERVENTIONS:
Procedure: Robotic gastric bypass with or without cholecystectomy — Study Arm: robotic gastric bypass without cholecystectomy Control Arm: robotic gastric bypass with cholecystectomy

SUMMARY:
The main objective of this pilot study is to show feasibility to collect peri-operative and postoperative clinical data of the study group of gastric bypass without cholecystectomy compared with the control group of gastric bypass with cholecystectomy. Our hypothesis is that the approach without cholecystectomy would be superior in terms of a decrease of perioperative adverse events and postoperative complications, as well as lenght of operation, lenght of hospital stay, overall costs with a very low risk of biliary complication in the follow up. These findings could be helpful to build a baseline for a future randomized controlled multicenter study allowing significance of these results and help orientate surgeons towards best surgical care of the gallbladder with confirmed absence of stones in the obese patient undergoing gastric bypass.

DETAILED DESCRIPTION:
We suggest performing a prospective randomized pilot trial comparing RYGB without concomitant cholecystectomy with RYGB with concomitant cholecystectomy for patients with absence of gallstones in preoperative ultrasound. Patients with ultrasonographically confirmed gallstones in the gallbladder undergo concomitant cholecystectomy at time of RYGB and are excluded from the study.Patients who meet the inclusion criteria will be randomized according to a randomization list generated by the CRC of the University Hospital of Geneva. The randomization envelops will be opened by the study staff at the appropriate time prior to the scheduling of gastric bypass after subject selection. The randomization assignment insert will contain information specifying whether the cholecystectomy will be performed or not during gastric bypass procedure.

A total of 90 consecutive obese patients attending the Unit of Visceral Surgery of the University Hospital of Geneva who meet the criteria for bariatric surgery and where the preoperative ultrasound confirms absence of gallstones will be recruited for the study.

A prospective open randomized pilot study design will be used. At 6 follow-up visits (at discharge, 1 ,3 ,6 ,12 and 18 months post-surgery), patients will be evaluated.

This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP or ISO EN 14155 as wella s all national legal and regulatory requirements, the LPth (Loi sur les produits thérapeutiques 812.21) and the OClin (Ordonnance sur les essais cliniques des produits thérapeutiques 812.214.2).

Description of surgical technique One optical trocar, three 12 mm trocars and one 5 mm trocar are placed. No additional trocar has to be placed for concomitant cholecystectomy. The intervention will start with the cholecystectomy laparoscopically. A small gastric pouch (around 20-30 cc) is created using blue cartridge staplers. A standard robotic RYGB with a 75 cm biliary limb and a 150 cm antecolic alimentary limb is performed. A hand-sewn gastrojejunal and jejunojejunal anastomois are performed, using a single layer running suture of Vicryl 2.0.

Data Collection:

Pre-Operative demographic data and other variables will be collected at baseline and at some of the 6 follow-up points (at discharge, 1,3,6,12,18 months):

Ultrasound, Patient Demographics and pre-Operative History will be collected, including: Gender, age on admission for operation, BMI, Height, Weight, ASA score, history of abdominal surgery, co- morbidities (Type 2 diabetes requiring Insulin or oral medication), Hypertension requiring medication, Coronary heart disease, including history of myocardial infarction, angina pectoris, coronary artery surgery Pulmonary comorbidities including history of pulmonary embolism, Sleep Apnea Tobacco use, Medication used by patient, Systolic and diastolic blood pressure, heart rate, Fasting plasma glucose, HbA1c, laboratory findings, QOL using the EQ-5D-5L questionnaire

Intra-Operative Assessment: Intra-Operative data such as complications (organ lesion, bleeding, conversion), operative time, docking times, estimated blood loss will be collected

Post-Operative Assessment: From surgery to discharge, the following patient information will be collected: complications according to Clavien/Dindo Classification system, re- operation, re-admission, length of hospital stay

Our hypothesis is that the approach without cholecystectomy would be superior in terms of a decrease of perioperative adverse events and postoperative complications, as well as lenght of operation, lenght of hospital stay, overall costs with a very low risk of biliary complication in the follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the criteria of the Swiss society for the study of morbid obesity (SMOB) to undergo gastric bypass (19):

  * BMI ≥ 35 kg/m2
  * Having followed a 2 year adequate program of weight loss without success or a 1 year program in case of "superobesity" (BMI ≥ 50 kg/m2)
  * Consent to multidisciplinary follow up for 5 years
* Preoperative ultrasound without presence of gallstones or polyps
* Age ≥ 18 years

Exclusion Criteria:

* Patients which have a contra-indication for gastric bypass according to the criteria of the Swiss society for the study of morbid obesity (SMOB) to undergo gastric bypass (19):

  * Pregnancy
  * Kidney failure (creatinine ≥ 300mmol/l, GFR < 30ml/min) without dialysis
  * Cirrhosis Child B/C
  * Ulcerative Colitis
  * Pulmonary embolism or deep venous thrombosis during the last 6 months
  * Psychiatric contra indications
  * Drug abuse (alcohol, cannabis, opioids) during the last 6 months
* Presence of gallstones on preoperative Ultrasound (which will require concomitant cholecystectomy)
* Patients with clinical diagnosis of cholecystitis defined as right upper quadrant abdominal pain, radiological signs of cholecystits and laboratory signs of infection or gallstone migration, defined as right upper quadrant and abnormal liver function tests (any increase in AST, ALT, alkaline Phosphatase, GGT and/or bilirubin).
* Previous bariatric surgery other than gastric banding
* Open bypass procedure
* Medical conditions preventing informed consent

Preoperative routine work-up includes a physical examination, vital parameters, laboratory analyses (hematology, chemistry and HbA1c), sleep apnea evaluation with Polygraphia, abdominal ultrasound, endoscopy of the stomach, pulmonary function, preoperative anesthesia consultation and psychological evaluation.

The results of these routine tests will be used to assess the patients'eligiibility to participate to the proposed pilot study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint consisting of: a.: intraoperative adverse events b.: postoperative complications | within 30 days after intervention
  Primary endpoint:
  1. composite endpoint consisting of:
  1. : intraoperative adverse events (common bile duct lesion, lesion of liver, lesion of digestive tract, bleeding, conversion).
  2. : postoperative complications according to Dindo/Clavien Classification

SECONDARY OUTCOMES:
Intraoperative adverse events in detail | day of operation
  * - Common bile duct lesion
  * - Lesion of Liver
  * - Lesion of digestive tract
  * - bleeding
  * - conversion
2. Morbidity and mortality | 18 months
  2. Morbidity and mortality assessed by Dindo/ Clavien Classification system
operation time | day of operation
  length of operation time
hospital stay | 6 months
  length of hospital stay (discharge criteria defined as follows : absence of fever (T≤37.8), Neutrophils ≤12G/L, Absence of anemia, no nausea, no vomiting)
gallstones | 18 months
  occurence of asymptomatic or symptomatic gallstones
biliary complication | 18 months
  cholecystitis, choledocholithiasis, cholangitis, biliary pancreatitis
cost | 18 months
  average cost
EQ-5D-5L | 12 months
  Quality of life using the EQ-5D-5L questionnaire
Readmission | 18 months
  Readmission
Re intervention | 18 months
  Re intervention (Cholecystectomy, transgastric ERCP, biliary Revision)

CONTACTS AND LOCATIONS:
Overall Officials: Minoa Jung, Dr, Principal Investigator — Visceral Surgery, Department of Surgery, University Hospital of Geneva
Locations (1):
- Visceral Surgery, Department of Surgery, University Hospital Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mason EE, Renquist KE. Gallbladder management in obesity surgery. Obes Surg. 2002 Apr;12(2):222-9. doi: 10.1381/096089202762552395. PMID 11975217
- [Result] Schmidt JH, Hocking MP, Rout WR, Woodward ER. The case for prophylactic cholecystectomy concomitant with gastric restriction for morbid obesity. Am Surg. 1988 May;54(5):269-72. PMID 3364862
- [Result] Shiffman ML, Sugerman HJ, Kellum JM, Brewer WH, Moore EW. Gallstone formation after rapid weight loss: a prospective study in patients undergoing gastric bypass surgery for treatment of morbid obesity. Am J Gastroenterol. 1991 Aug;86(8):1000-5. PMID 1858735
- [Result] Everhart JE. Contributions of obesity and weight loss to gallstone disease. Ann Intern Med. 1993 Nov 15;119(10):1029-35. doi: 10.7326/0003-4819-119-10-199311150-00010. PMID 8214980
- [Result] Worni M, Guller U, Shah A, Gandhi M, Shah J, Rajgor D, Pietrobon R, Jacobs DO, Ostbye T. Cholecystectomy concomitant with laparoscopic gastric bypass: a trend analysis of the nationwide inpatient sample from 2001 to 2008. Obes Surg. 2012 Feb;22(2):220-9. doi: 10.1007/s11695-011-0575-y. PMID 22183984
- [Result] Patel KR, White SC, Tejirian T, Han SH, Russell D, Vira D, Liao L, Patel KB, Gracia C, Haigh P, Dutson E, Mehran A. Gallbladder management during laparoscopic Roux-en-Y gastric bypass surgery: routine preoperative screening for gallstones and postoperative prophylactic medical treatment are not necessary. Am Surg. 2006 Oct;72(10):857-61. PMID 17058721
- [Result] Weinsier RL, Ullmann DO. Gallstone formation and weight loss. Obes Res. 1993 Jan;1(1):51-6. doi: 10.1002/j.1550-8528.1993.tb00008.x. PMID 16350561
- [Result] Wudel LJ Jr, Wright JK, Debelak JP, Allos TM, Shyr Y, Chapman WC. Prevention of gallstone formation in morbidly obese patients undergoing rapid weight loss: results of a randomized controlled pilot study. J Surg Res. 2002 Jan;102(1):50-6. doi: 10.1006/jsre.2001.6322. PMID 11792152
- [Result] Warschkow R, Tarantino I, Ukegjini K, Beutner U, Guller U, Schmied BM, Muller SA, Schultes B, Thurnheer M. Concomitant cholecystectomy during laparoscopic Roux-en-Y gastric bypass in obese patients is not justified: a meta-analysis. Obes Surg. 2013 Mar;23(3):397-407. doi: 10.1007/s11695-012-0852-4. PMID 23315094
- [Result] Villegas L, Schneider B, Provost D, Chang C, Scott D, Sims T, Hill L, Hynan L, Jones D. Is routine cholecystectomy required during laparoscopic gastric bypass? Obes Surg. 2004 Jan;14(1):60-6. doi: 10.1381/096089204772787301. PMID 14980035
- [Result] Tucker ON, Fajnwaks P, Szomstein S, Rosenthal RJ. Is concomitant cholecystectomy necessary in obese patients undergoing laparoscopic gastric bypass surgery? Surg Endosc. 2008 Nov;22(11):2450-4. doi: 10.1007/s00464-008-9769-3. Epub 2008 Feb 21. PMID 18288531
- [Result] Buchs NC, Morel P, Azagury DE, Jung M, Chassot G, Huber O, Hagen ME, Pugin F. Laparoscopic versus robotic Roux-en-Y gastric bypass: lessons and long-term follow-up learned from a large prospective monocentric study. Obes Surg. 2014 Dec;24(12):2031-9. doi: 10.1007/s11695-014-1335-6. PMID 24962109